CLINICAL TRIAL: NCT00759798
Title: Prospective Identification of Significant Prognostic Factors in Patients Treated With Fludarabine, Cyclophosphamide, and Rituximab (FCR) as Initial Therapy for Chronic Lymphocytic Leukemia.
Brief Title: Identifying Prognostic Factors in Frontline FCR for Patients With Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0431; NCI-2012-01663 (Registry Identifier: NCI CTRP); 246915 (Other Grant/Funding Number: Evaluation of Biomarkers for CLL Progression in the p53 Pathway: A Genetic Approach in Mice and Man)
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Chronic Lymphocytic Leukemia; Leukemia
Keywords: Chronic Lymphocytic Leukemia; Leukemia; FCR; Fludarabine; Cyclophosphamide; Rituximab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fludarabine, Cyclophosphamide, Rituximab (Experimental): Fludarabine 25 mg/m^2 given intravenously on Days 2-4 of Cycle 1 and Days 1-3 of Cycles 2 and beyond. Cyclophosphamide 250 mg/m2 given intravenously on Days 2-4 of Cycle 1 and Days 1-3 of Cycles 2 and beyond. Rituximab 375 mg/m2 given intravenously on Day 1 of Course 1
  All subsequent Courses: 500 mg/m2 given intravenously on Day 1 (Weeks 5,9,13,17,21)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Rituximab

INTERVENTIONS:
Drug: Fludarabine — 25 mg/m^2 given intravenously on Days 2-4 of Cycle 1 and Days 1-3 of Cycles 2 and beyond.
  Other Names: Fludara®
Drug: Cyclophosphamide — 250 mg/m2 given intravenously on Days 2-4 of Cycle 1 and Days 1-3 of Cycles 2 and beyond.
  Other Names: Cytoxan®; Neosar®
Drug: Rituximab — 375 mg/m2 given intravenously on Day 1 of Course 1
  All subsequent Courses: 500 mg/m2 given intravenously on Day 1 (Weeks 5,9,13,17,21)
  Other Names: Rituxan®

SUMMARY:
The goal of this clinical research study is to learn more about the characteristics of CLL, including genes and chromosome abnormalities and proteins expressed by the leukemia cells, which may help doctors predict if patients who receive standard treatment (fludarabine, cyclophosphamide, and rituximab) for the first time will experience a complete remission.

DETAILED DESCRIPTION:
The Study Drugs:

Fludarabine is designed to make cancer cells less able to repair damaged DNA (the genetic material of cells). This may increase the likelihood of the cells dying.

Cyclophosphamide is designed to interfere with the multiplication of cancer cells, which may slow or stop their growth and spread throughout the body. This may cause the cancer cells to die.

Rituximab is designed to attach to lymphoma cells, which may cause them to die.

Study Drug Administration:

Each cycle is 4-6 weeks.

If you are found to be eligible to take part in this study, on Day 1 of each cycle, you will receive rituximab through a needle into your vein over 6-8 hours.

On Days 2-4 of Cycle 1 and Days 1-3 of Cycles 2 and beyond, you will receive fludarabine by vein over 30 minutes. You will also receive cyclophosphamide by vein over 30 minutes.

You will receive drugs (such as Tylenol, Benadryl, Zofran, allopurinol, and Valtrex) to help prevent side effects. If you have side effects while receiving rituximab, you may be monitored by the study staff for 2 hours after each dose.

Study Visits:

Once a week, blood (about 1 tablespoon) will be drawn for routine tests.

After 3 months (3 cycles of treatment), the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will have a bone marrow aspirate and biopsy to check the status of the disease.

Length of Study:

You will be on treatment for about 6 months. You will be taken off treatment early if you have intolerable side effects or the disease gets worse.

End-of-Treatment Visit:

After you are off treatment, you will have an end-of-treatment visit for doctors to learn your overall response to the treatment. The following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will have a bone marrow aspirate and biopsy to check the status of the disease.

Long-Term Follow-up:

At 6 months after you have finished treatment and then every year from then on, you will have follow-up visits. The following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* If your doctor thinks it is needed, you will have a bone marrow biopsy and aspirate to check the status of the disease.

This is an investigational study. Fludarabine, cyclophosphamide, and rituximab are FDA approved and commercially available for the treatment of CLL. The correlation with response to treatment and the characteristics of the leukemia cells is investigational.

Up to 300 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will have a diagnosis of CLL, Small Lymphocytic Lymphoma (SLL), or CD20 positive low-grade lymphoproliferative disorder.
2. All patients with untreated Rai stage III-IV are eligible for this protocol. Prior treatment with single-agent rituximab permitted. OR Patients with untreated Rai stage 0-II who meet one or more criteria for active disease as defined by the International Working Group for CLL (IWCLL). Prior treatment with single-agent rituximab permitted.
3. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3.
4. Patients must have adequate renal and hepatic function (creatinine <2mg%, bilirubin <2mg%). Patients with renal or liver dysfunction due to organ infiltration by lymphocytes may be eligible after discussion with the study chairman.
5. Patients may not receive other concurrent chemotherapy, radiotherapy, or immunotherapy. Localized radiotherapy to an area not compromising bone marrow function does not apply.
6. Patients must be 16 years of age or older.
7. Patients must sign informed consent indicating that they are aware of the investigational nature of this study according to the policies of the MD Anderson Cancer Center Institutional Review Board (MDACC IRB).

Exclusion Criteria:

N/A

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2008-08-13 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Wierda, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Strati P, Keating MJ, O'Brien SM, Burger J, Ferrajoli A, Jain N, Tambaro FP, Estrov Z, Jorgensen J, Challagundla P, Faderl SH, Wierda WG. Eradication of bone marrow minimal residual disease may prompt early treatment discontinuation in CLL. Blood. 2014 Jun 12;123(24):3727-32. doi: 10.1182/blood-2013-11-538116. Epub 2014 Apr 4. PMID 24705492
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 2008 to April 2016
Groups:
- Fludarabine, Cyclophosphamide, Rituximab: Fludarabine 25 mg/m^2 given intravenously on Days 2-4 of Cycle 1 and Days 1-3 of Cycles 2 and beyond. Cyclophosphamide 250 mg/m2 given intravenously on Days 2-4 of Cycle 1 and Days 1-3 of Cycles 2 and beyond. Rituximab 375 mg/m2 given intravenously on Day 1 of Course 1
  All subsequent Courses: 500 mg/m2 given intravenously on Day 1 (Weeks 5,9,13,17,21)
  Fludarabine: 25 mg/m^2 given intravenously on Days 2-4 of Cycle 1 and Days 1-3 of Cycles 2 and beyond.
  Cyclophosphamide: 250 mg/m2 given intravenously on Days 2-4 of Cycle 1 and Days 1-3 of Cycles 2 and beyond.
  Rituximab: 375 mg/m2 given intravenously on Day 1 of Course 1
  All subsequent Courses: 500 mg/m2 given intravenously on Day 1 (Weeks 5,9,13,17,21)
Period: Overall Study
Arm/Group | Fludarabine, Cyclophosphamide, Rituximab
Started | 289
Completed | 289
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fludarabine, Cyclophosphamide, Rituximab
Number analyzed (Participants) | 289
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 237
  >=65 years | 52
Age, Continuous [Median (Full Range); unit: years] | 59 [32 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 183
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 256
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 289

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Remission (CR)
Description: Complete Response defined by NCI Working Group / International Working Group for CLL criteria as no evidence of disease on physical examination (no adenopathy or organomegaly) or microscopic examination of blood (ALC <4,000/L) and bone marrow (<30% lymphocytes, no lymphoid nodules), and recovery of hemoglobin, neutrophil, and platelet counts.
Time Frame: After 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fludarabine, Cyclophosphamide, Rituximab
Number analyzed (Participants) | 289
Participants | 185

ADVERSE EVENTS:
Time Frame: Up to 7 years, 8 months
Arm/Group | Fludarabine, Cyclophosphamide, Rituximab
All-Cause Mortality (participants affected / at risk) | 20/289
Serious Adverse Events (participants affected / at risk) | 65/289
Other Adverse Events (participants affected / at risk) | 0/289
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fludarabine, Cyclophosphamide, Rituximab (N=289)
Fever (General disorders) | 15 (18)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Neutropenic Fever (Blood and lymphatic system disorders) | 22 (23)
Infection (Infections and infestations) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Abdominal Pain (General disorders) | 3 (3)
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 8 (12)
Nausea/Vomiting (Gastrointestinal disorders) | 1 (1)
Hyperbilirubinemia (Investigations) | 1 (2)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Perineal Abcess (Reproductive system and breast disorders) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1)
staphylococcus Infection Leg (Infections and infestations) | 1 (1)
Opportunistic Infection (Infections and infestations) | 2 (2)
Pain Lower Extremity (General disorders) | 1 (1)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Flu Like Symptoms (General disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT00759798/Prot_SAP_000.pdf